CLINICAL TRIAL: NCT05359783
Title: Sentinel Node Localization and Staging with Low Dose Superparamagnetic Iron Oxide-enhanced Magnetic Resonance Imaging and Magnetic Probe in Patients with Breast Cancer
Brief Title: Sentinel Node Localization and Staging with Low Dose Superparamagnetic Iron Oxide
Acronym: MAGSNOW
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Principal investigator, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUGBG-2021001
Record Dates: First submitted 2022-04-06; First posted 2022-05-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: Breast cancer; Sentinel Lymph Node Biopsy; Superparamagnetic iron oxide
MeSH Terms: conditions — Breast Neoplasms | interventions — ferumoxides

STUDY DESIGN:
Intervention Model Description: A phase Ib/II interventional dose-escalation single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentinel node detection with 0.1mL SPIO (Experimental): An intradermal injection of SPIO (MagTrace®), according to the pre-specified dose of 0.1mL, will be performed 7 days, up to the day of surgery. The injection should be in the skin over the tumour, or at the border of the areola
  Interventions: Drug: Superparamagnetic Iron Oxide

INTERVENTIONS:
Drug: Superparamagnetic Iron Oxide — Superparamagnetic iron oxide (SPIO) consists of an iron oxide nanoparticle core and a hydrophilic coating to make it biocompatible and colloidal stable in a suspension.
  Other Names: MagTrace

SUMMARY:
Sentinel lymph node (SLN) status is pivotal for treatment decisions in breast cancer patients. The dual technique with Technetium99m (Tc99) and blue dye (BD) is yet the current routine for SLN detection. However, the same reliability has been presented by superparamagnetic iron oxide nanoparticles (SPIO). The aim of this study was to determine if SLN detection using ultra-low dose SPIO is feasible.

DETAILED DESCRIPTION:
Sentinel lymph node (SLN) status is pivotal for treatment decisions in breast cancer patients. The dual technique with Technetium99m (Tc99) and blue dye (BD) is yet the current routine for SLN detection. However, the same reliability has been presented by superparamagnetic iron oxide nanoparticles (SPIO). The aim of this study was to determine if SLN detection using ultra-low dose SPIO is feasible.

This is a phase Ib/II interventional dose-escalation single arm study. There will be a dose escalation of SPIO (0.1ml, 0.25ml and 0.5 ml) with a minimum of 5 patients per step. If 4 or more procedures are successful, no further dose escalation will be performed. 30 patients will be included with the minimal successful dose.

Furthermore, a total of 20 patients with the minimal successful dose will be included for the secondary objective A - to evaluate if it is possible to map and stage sentinel lymph nodes with SPIO-enhanced axillary MRI. For the secondary objective B - an additional of 20 patients with the minimal successful dose will be included to evaluate if SPIO in a low dose creates any SPIO related artifacts on breast MRI after breast conserving surgery. These two parts of the study are optional, and the patients will be asked specifically about participation in these two objectives, A and B. All included patients will be evaluated for skin staining at study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged above 18 years
2. Signed and dated written informed consent before the start of specific protocol procedures
3. Histologically confirmed breast cancer planned for breast conserving surgery and sentinel lymph node biopsy

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Iron overload disease
3. Known hypersensitivity to iron, dextran compounds or blue dye.
4. Inability to understand given information and give informed consent or undergo study procedures
5. MRI (subgroup of patients): Conditions contraindicating MRI including, but not limited to, BMI > 40 kg/m2, claustrophobia, metallic implants or internal electrical devices (e.g., pacemaker) and permanent makeup or tattoos which in the Investigator's opinion might jeopardise the patient's safety or imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node detection rate compared to Tc99m and blue dye | During the procedure
  To evaluate the use of superparamagnetic iron oxide (SPIO) as a tracer in a minimal lower dose (0.1-0.5 ml) for sentinel lymph node detection in breast cancer.

SECONDARY OUTCOMES:
MRI artefacts in breast | 6 and 12 months after surgery
  To evaluate if SPIO in a low dose creates any SPIO related breast MRI artefacts (assessed by breast MRI), reported as percentage of patients with artefacts present.
SPIO related skin staining | 6 and 12 months after surgery
  To evaluate if SPIO in a low dose creates any SPIO related skin staining (assessed by photo), reported as percentage of patients with artefacts present.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waanders S, Visscher M, Wildeboer RR, Oderkerk TO, Krooshoop HJ, Ten Haken B. A handheld SPIO-based sentinel lymph node mapping device using differential magnetometry. Phys Med Biol. 2016 Nov 21;61(22):8120-8134. doi: 10.1088/0031-9155/61/22/8120. Epub 2016 Oct 26. PMID 27782005
- [Background] Karakatsanis A, Daskalakis K, Stalberg P, Olofsson H, Andersson Y, Eriksson S, Bergkvist L, Warnberg F. Superparamagnetic iron oxide nanoparticles as the sole method for sentinel node biopsy detection in patients with breast cancer. Br J Surg. 2017 Nov;104(12):1675-1685. doi: 10.1002/bjs.10606. Epub 2017 Sep 6. PMID 28877348
- [Background] Karakatsanis A, Christiansen PM, Fischer L, Hedin C, Pistioli L, Sund M, Rasmussen NR, Jornsgard H, Tegnelius D, Eriksson S, Daskalakis K, Warnberg F, Markopoulos CJ, Bergkvist L. The Nordic SentiMag trial: a comparison of super paramagnetic iron oxide (SPIO) nanoparticles versus Tc(99) and patent blue in the detection of sentinel node (SN) in patients with breast cancer and a meta-analysis of earlier studies. Breast Cancer Res Treat. 2016 Jun;157(2):281-294. doi: 10.1007/s10549-016-3809-9. Epub 2016 Apr 27. PMID 27117158
- [Background] Motomura K, Izumi T, Tateishi S, Sumino H, Noguchi A, Horinouchi T, Nakanishi K. Correlation between the area of high-signal intensity on SPIO-enhanced MR imaging and the pathologic size of sentinel node metastases in breast cancer patients with positive sentinel nodes. BMC Med Imaging. 2013 Sep 13;13:32. doi: 10.1186/1471-2342-13-32. PMID 24028426
- [Background] Motomura K, Izumi T, Tateishi S, Tamaki Y, Ito Y, Horinouchi T, Nakanishi K. Superparamagnetic iron oxide-enhanced MRI at 3 T for accurate axillary staging in breast cancer. Br J Surg. 2016 Jan;103(1):60-9. doi: 10.1002/bjs.10040. Epub 2015 Nov 17. PMID 26572241
- [Background] Jazrawi A, Pantiora E, Abdsaleh S, Bacovia DV, Eriksson S, Leonhardt H, Warnberg F, Karakatsanis A. Magnetic-Guided Axillary UltraSound (MagUS) Sentinel Lymph Node Biopsy and Mapping in Patients with Early Breast Cancer. A Phase 2, Single-Arm Prospective Clinical Trial. Cancers (Basel). 2021 Aug 25;13(17):4285. doi: 10.3390/cancers13174285. PMID 34503095